CLINICAL TRIAL: NCT02356536
Title: The Effect of a Wearable Cueing Device on Freezing of Gait in Parkinson's Disease
Acronym: CuePed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, rodney marsh, Dr, The University of Queensland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013000952
Record Dates: First submitted 2015-01-28; First posted 2015-02-05 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Gait Disorders, Neurologic
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Device: Agilitas

INTERVENTIONS:
Device: Agilitas — WCD trial

SUMMARY:
The CuePeD trial is an intervention trial measuring the effectiveness of a novel treatment for Freezing of Gait (FOG) in Parkinson's disease (PD). The primary intervention is the use of a wearable cueing device (WCD), which detects and responds to FOG and extinguishes on the resumption of normal walking. It is designed for use in PD patients with FOG, in their home environment where FOG is most severe. Kinematic data will be logged by a memory card in the belt worn device recording FOG, and falls. The device will be used on 3 different settings in a gait laboratory environment, and then for 2 weeks in the patient's own home using the same 3 settings. A battery of psychometric instruments will be administered before and after the trial

DETAILED DESCRIPTION:
The CuePeD trial primarily involves the use of a WCD ( pictured on website www.brightdevices.com.au). This is a belt worn device, with a co-location of motion sensor input and cueing output. The input is mediated by miniaturized accelerometers and gyroscopes and utilizes software algorithms which have been developed to detect FOG. The cueing output is mediated by a laser light which shines on the floor in front of the user as a continuous visual signal. The cue is produced because of the device's ability to recognize FOG in the user. The laser is produced for a predetermined period of time or until normal gait is recommenced, at which time it extinguishes until the next freezing episode.

This study plans to examine the effectiveness of the WCD for the problem of FOG in PD 'in vivo', that is, in a community setting.

FOG has been defined narrowly as 'the sudden inability to initiate or sustain locomotion'. It includes 'start', 'turn' and 'destination' hesitation. A broader definition accepted at the 2010 workshop of clinicians and scientists interested in FOG was " brief, episodic absence or marked reduction of forward progression of the feet despite the intention to walk" . It generally occurs several years after the onset of PD and has been recognized as a significant source of morbidity in PD patients. Cueing represents one of the more promising treatments, but the demonstration of in vivo effectiveness of this intervention to date, are modest.

Falls, while often multifactorial in a general population, in PD are often attributable to FOG.

Unfortunately, current treatments for FOG are largely ineffective, and the evidence for their use limited.

Interventions for FOG are usually pharmacological and involve manipulation of laevodopa (LD) doses, or more recently, the addition of stimulants. Other centrally acting medications have been described anecdotally as beneficial, but have not been systematically studied.

Possibly as a consequence of the decrease in postoperative laevodopa (LD) dose in chronic users, or the under recognized significance of the subthalamic nucleus ( the most common stimulation target) in gait regulation, the rise of Deep Brain Stimulation as a treatment for PD may contribute to the problem.

The first study employing a wearable device to detect FOG was described by Bachlin in 2010, but involved a 3 component device (an ankle worn motion sensor, belt worn processing unit and earpiece for cueing output) and a pulsed auditory cue (a 1 Hz clicking sound).

One of the recurring difficulties for gait scientists is the inability to elicit FOG in freezers' in vitro' in the laboratory. This is due to the artificial clinical environment giving rise to a 'best performance' or 'paradoxical kinesia'.

Non-laboratory, 'in vivo' measures have been limited to user rated questionnaires at the end of a trial period of in home use.

This freeze detecting, cue producing device offers an elegant solution for the amelioration of FOG and possibly falls in a PD population in their day to day life. In addition, it offers a novel opportunity for the objective measurement of kinematic data to assess the efficacy of the device in individual subjects.

Whilst cueing has been recognized as a treatment for FOG for more than 25 years, most of this work has occurred in gait laboratories. It is well known that FOG is induced in many subjects with initiation of gait, turns and 'dual tasking'. This commonly occurs in the domestic environment, where there are small spaces doorways, hallways etc.

Most 'in vitro' work has taken place with a fixed, pulsed cue, usually auditory, but including visual and somatosensory/vibration pulses. Unfortunately, the landmark 2006 RESCUE trial of Neiubauer demonstrated an improvement in gait that was not sustained once the cueing device was removed. That is, the problem of FOG is not readily rehabilitated with cueing, and benefits of cueing training quickly extinguish once the treatment finishes.

The neurobiology of why FOG occurs in this setting, while beyond the scope of this description, is beginning to be understood, and is worthy of brief commentary to better understand the WCD's mechanism of action. Several lines of evidence, including functional imaging studies point to a failure of reconciliation of motor, cognitive and emotional circuits in FOG prone patients. Mental tasks (such as counting backwards), additional motor tasks (such as carrying a glass of water), as well as a feeling of severe anxiety itself can all induce FOG. The presence of a doorway or kitchen bench, which requires contemplation, similarly represents a dual tasking challenge which can induce FOG. Being optimally emotionally aroused in a laboratory setting can assist overcoming the propensity to freeze.

The proposed research will be a case series analysis of 30 PD patients with clinically significant FOG; recruited from local movement disorder neurologists. There will be no blinding. There will be an ABA design with subjects acting as their own controls - the device on continually, on during FOG episodes or off at different time periods. There will be randomization of the 3 device settings for different time periods.

Each trial will take 2 weeks, with an initial gait laboratory assessment. During this assessment signature freezing episodes will be captured, videoed, for each patient, and correlated with kinematic readings. identification of FOG episodes and Inter-rater reliability data will be obtained during these assessments. Patients will become familiar with the use of the device for later use at home. 3 tasks will be undertaken by each patient on each device setting - ie 9 tasks in total - these include: a timed up and go, 2 minute walk and a specifically designed obstacle course. A battery of psychometric instruments will be completed.

This assessment will then be followed by a 2 week home trial. 3 device settings will be employed in both environments - 1. the device 'off' and simply measuring FOG using its software algorithms, 2.the device "on" whereby FOG episodes trigger the laser cue, and 3. the device on 'continually' whereby, a continuous visual cue is emitted from the device, independent of FOG episodes .

The device will be on settings 1,2 and 3 for 3,7 and 4 days respectively, with randomisation of the order of settings 2 and 3.

During the 2 week home trial, Kinematic data to capture FOG duration will be logged on the device during the same time period each day with the device on different settings. Fall data will collected from 6am to 10pm.

Crucially, FOG episodes on all 3 settings of the device will be recorded. The primary outcome measure will be the total seconds of FOG when the device is simply recording compared with the total FOG seconds when a FOG dependent ( or continuous FOG independent) cue is provided by the device.

At the end of the 7 days on setting 2 (FOG dependent cue), instrument ratings will be completed for a second time, and returned with the device for collation of the data.

Whilst cueing has been recognized as a treatment for FOG for more than 25years, most of this work has occurred in gait laboratories. It is well known that FOG is induced in many subjects with initiation of gait, turns and 'dual tasking'. This commonly occurs in the domestic environment, where there are small spaces doorways, hallways etc.

One hypothesis regarding the limited efficacy conferred by current devices used for FOG, is that pulsed, fixed auditory stimuli represent a cognitive burden and may actually induce FOG once the initial freeze is overcome. The work of Wolpert would suggest that a pulsed auditory cue extending beyond the freezing episode would at best be 'gated' out by the subject, and essentially ignored. Bachlin's subjects complained that the auditory cue was annoying.

A fixed visual cue which extinguishes after the freeze is broken appeals as a powerful antidote to this paradox of focusing the patient's attention at the point of freezing, but not adding to their cognitive burden once the freeze is broken. This was recognized with the first descriptions of cueing for FOG with an inverted walking cane. It is a powerful example of the curiosity of paradoxical kinesia well known to the disorder, and not easily forgotten by clinicians who have been witness to it. Until the recent development of increasingly miniaturized, sophisticated accelerometers and gyroscopes, there was no mechanism to replicate the effect of an upturned cane held by a walking companion.

It is now known that there is an increasing loss of automaticity in FOG patients, and an increase in cortical connectivity with deep brain structures - that is, there seems to be a 'cortical takeover' of gait in these patients. It seems likely that a cue may more readily enable a re-accessing of 'vestigial' gait motor programs in those patients that it helps.

The 2 null hypotheses of the research project will be: (1)That the wearable, freeze detecting cueing device has no measurable effect on total freeze duration, total number of freezing episodes , or total number of falls over the same three 1 hour intervals measured on separate days in subjects with Parkinson's disease; and:(2)That there is no difference in user rated instrument measures of Quality of Life, Freezing of Gait, Falls, Anxiety and Depression before and after 2 weeks of treatment a wearable, freeze detecting cueing device in patients with Parkinson's disease.

The proposed research will be a case series analysis of 30 PD patients with clinically significant FOG; recruited from local movement disorder neurologists. There will be no blinding. In both arms of the trial, there will be an ABA design with subjects acting as their own controls - the device on and off at different time periods.

The assessments will include:

1. Freezing of Gait Questionnaire(FOGQ); Falls Efficacy Scale (FES); Parkinson's Disease Questionnaire 39; Geriatric Anxiety Inventory (GAI), Geriatric depression scale (GDS); Spielberger Trait Anxiety Inventory (STAI); Mini mental state examination MMSE and MOCA .
2. 2minute walk test; Timed 'up and go' test; Dual tasking Timed up and go test; standardized 20 metre obstacle course that includes a doorway, corridor, 180 and 360 degree turns.

Patients will then be asked to take the WCD home for 14 days with clear guidelines for its use. The battery of questionnaires to be completed at the end of the 14 days, along with a self addressed postal pack for the return of the device will accompany the patient.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's Disease, clinically significant freezing of gait, no significant medical comorbidities

Exclusion Criteria:

* Non-english speaking, dementia, wheelchair or mobility aid dependent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Total seconds of FOG | 2 weeks
  duration of freezing with device on versus During the 2 week home trial, Kinematic data to capture FOG duration will be logged on the device during the same time period each day with the device on different settings. Fall data will collected from 6am to 10pm.
  FOG episodes on all 3 settings of the device will be recorded. The primary outcome measure will be the total seconds of FOG when the device is simply recording compared with the total FOG seconds when a FOG dependent ( or continuous FOG independent) cue is provided by the device. This will be recorded by means of a microSD card within the device. The data will be downloaded once the device is returned

CONTACTS AND LOCATIONS:
Overall Officials: rodney i marsh, MBBS, Principal Investigator — The University of Queensland
Locations (1):
- University of Queensland, Brisbane, Queensland, Australia